CLINICAL TRIAL: NCT06568224
Title: Treatment for Hidradenitis Suppurativa
Brief Title: Therapeutic Effect of Methalazine on 27 Cases of Suppurative Hidradenitis
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hou Maihua, Chief physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: HouMaihua
Record Dates: First submitted 2024-05-27; First posted 2024-08-23 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Mesalamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mesalazine — oral mesalazine 1g qid

SUMMARY:
Background: Hidradenitis suppurativa (HS) is a chronic inflammatory relapsing disease involving the axillae, breast ,groin and anogenital regions. The therapies of the disease are diverse, including medication and surgery. However, responses to treatments are variable and relapse is common, with no single agent being consistently effective.

Objective: To evaluate the efficacy and safety of oral mesalazine treatment for hidradenitis suppurativa .

Methods: Investigators reported a series of cases of patients who received oral mesalazine(1g qid) for hidradenitis suppurativa in our institution between May 2020 and September 2023. A total of 27 patients, 22 in the mild to moderate group and 5 in the severe group, were included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent painful or suppurative lesions
* Typical clinical manifestations: the distribution of apocrine sweat glands is deep in painful nodules, abscesses, sinuses, scars;

Exclusion Criteria:

* Severe neurological and psychiatric diseases
* Tumor diseases
* Pregnant women in lactation period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The symptoms of the patients were papules, nodules, cysts, sinuses, pustules, fistulas and scars in the armpits, groin, buttocks, etc., often accompanied by significant pain and tenderness.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic Effect of Methalazine on 27 Cases of Suppurative Hidradenitis | Three and a half years
  We registered the number of patients who achieved HiSCR（%）.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT06568224/Prot_SAP_001.pdf